CLINICAL TRIAL: NCT01256112
Title: Parent Supported Weight Reduction in Down Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: University of Massachusetts, Worcester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1 R03 DK070627 (completed); R03DK070627 (NIH)
Record Dates: First submitted 2010-12-06; First posted 2010-12-08 (Estimated); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Down Syndrome
Keywords: obesity; behavioral intervention; family based; weight loss
MeSH Terms: conditions — Down Syndrome; Obesity; Weight Loss | interventions — Behavior Therapy; Nutritional Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NAE + Behavioral Intervention (Experimental): Parents of participants receive training in behavioral support at home, in addition to a standard nutrition and physical activity education (NAE) program.
  Interventions: Behavioral: Parent Supported Behavioral Intervention; Behavioral: Nutrition/Activity Education (NAE)
- Nutrition/Activity Education (Active Comparator): Parents and participants receive a standard nutrition and physical activity education (NAE) program.
  Interventions: Behavioral: Nutrition/Activity Education (NAE)

INTERVENTIONS:
Behavioral: Parent Supported Behavioral Intervention — Parents of participants receive training in behavioral support at home in order to facilitate lifestyle change associated with dietary choices and physical activity designed to produce gradual weight loss.
  Other Names: lifestyle modification; behavior modification; behavior therapy
  Arms: NAE + Behavioral Intervention
Behavioral: Nutrition/Activity Education (NAE)

SUMMARY:
The purpose of this study is to determine whether a nutrition and physical activity education program for families of overweight or obese adolescents with Down syndrome is more effective when behavioral lifestyle change strategies are added.

DETAILED DESCRIPTION:
Children with intellectual disabilities, including Down syndrome (DS), are as likely to be overweight than their typically developing peers. The consequences of childhood obesity include increased risk for Type-2 diabetes, orthopedic problems, sleep apnea, elevated cardiovascular risk and menstrual irregularities. Research indicating a high prevalence of overweight, obesity, low fitness levels and other health problems among adults with DS suggest the need for more attention to health promotion among adolescents with DS, which has been limited to date. Educational interventions in nutrition and physical activity have not been tested through randomized clinical trial with families of adolescents with DS; nor have behavioral "lifestyle change" interventions based on Social Cognitive Theory. Among typical populations, the addition of training in behavior and lifestyle change to education-alone interventions increasingly is being seen as critical in helping to promote long-term weight loss and weight maintenance. The hypothesis of this study is that a parent supported weight reduction (PSWR) intervention that combines behavioral strategies with nutrition and activity education (NAE) will be more effective in reducing overweight in adolescents with DS than a program that provides NAE alone or a Wait-List (WL) control.

ELIGIBILITY:
Inclusion Criteria:

* Age 13-26 with Down syndrome
* Living at home in single- or two-parent family, w/no plans to leave home in next year
* Achieves IQ score 45 or above on the Kaufman Brief Intelligence Test (K-BIT)
* Academic ability and necessary behavioral/social control to participate in a group classroom-based educational program
* Clinically overweight, as indicated by a BMI at or above 85th percentile for age and gender
* Signed approval to participate, which includes a completed recent thyroid screen, provided by participant's Primary Physician (and participant's cardiologist is he/she has a history of a heart condition), and participant's neurologist if he/she has a history of seizures)

Exclusion Criteria:

* Untreated thyroid disorder
* Type I or II Diabetes
* Cardiac problem, treated or untreated, for whom the participant's treating cardiologist indicates restrictions in physical activity
* Epilepsy/seizure disorder in which participant is not stable on medications
* Orthopedic injuries or deformities
* Chronic GI illness (except constipation) including inflammatory bowel diseases and celiac disease
* Prader Willi syndrome
* Unwillingness to wear accelerometer at screening or enrollment
* Non-ambulatory, i.e., uses wheelchair or other assistive devices for moving about and walking
* Chronic/severe foot infection (as screened by physical therapist, but in coordination with physician)
* Severe balance problems (as screened by physical therapist)
* Resting heart rate less than 50 beats per minute (bpm), or greater to or equal to 100 bpm (observed in physical therapy screening)
* History of major medical illness (i.e., cancer, leukemia)
* History of profound behavioral problems, i.e., self injury, injury to others, property destruction, etc.
* Other diagnosed disorders, including autism spectrum disorders, bipolar disorder (within the last year), eating disorder (within the last year), major depression (within the last year), psychosis & schizophrenia
* Other exclusion conditions left to the discretion of the study team

Ages: 13 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2006-09; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard K Fleming, PhD, Principal Investigator — University of Massachusetts Medical School, Eunice Kennedy Shriver Center
Locations (1):
- Eunice Kennedy Shriver Center at UMASS Medical School, Waltham, Massachusetts, United States

REFERENCES:
- [Result] Curtin C, Bandini LG, Must A, Gleason J, Lividini K, Phillips S, Eliasziw M, Maslin M, Fleming RK. Parent support improves weight loss in adolescents and young adults with Down syndrome. J Pediatr. 2013 Nov;163(5):1402-8.e1. doi: 10.1016/j.jpeds.2013.06.081. Epub 2013 Aug 20. PMID 23968742
- See also: Web site for organization in which research was conducted — http://www.umassmed.edu/shriver/index.aspx